CLINICAL TRIAL: NCT04975113
Title: The Effects of Progressive Neuromuscular Exercise Program and Taping on Muscle Strength and Pain in Patellofemoral Pain: A Randomized Controlled Blind Study
Brief Title: The Effects of Progressive Neuromuscular Exercise Program and Taping on Muscle Strength and Pain in Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 13/314-01
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Patellofemoral Pain Syndrome; Kinesiotape; Exercise; Strength
Keywords: strength; neuromuscular exercise; Kinesiotape; Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients were given a progressive neuromuscular exercise program that included stabilization of the knee and hip joint . Green color elastic band was used in resistant exercises. When subjects used the green color Thera-Band®, they started with an easy length and increased relative to the Omni Scale .
  Interventions: Other: progressive neuromuscular exercise program
- Exercise and Taping group (Experimental): Patients in this group received the same exercises given in the "exercise group" for 12 weeks. In addition to these exercises, mechanical correction tape (5cm, Kinesio Tex Gold®) was applied for the knee and foot.
  Interventions: Other: Exercise and Taping

INTERVENTIONS:
Other: progressive neuromuscular exercise program — The exercises to be performed in the following week at the beginning of each week were explained by the researcher physiotherapist on the brochure and given as a home program and continued for a total of 12 weeks. The researcher physiotherapist saw the patients every week and carried out exercise compliance and control.
  Arms: Exercise group
Other: Exercise and Taping — "I" taping for accurate positioning of the tissue was applied to the patients to neutralize the patellofemoral joint. During the knee flexion in the supine position, the tape was adhered to the skin with a moderate-to-extreme stretch (50%-75%) . Clinical therapeutic applications of the Kinesio taping methods (Tokyo, Japan: Ken Ikai Co Ltd.). In addition to the patellar taping, correction taping to neutralize the subtalar joint by elevating the midtarsal joint and medial arch was applied. The patients were positioned in prone lying and knee flexion position, the taping was started at the 5th metatarsal level on the dorsal side of the finger and finished extending towards the medial of the tibia . Tapings were renewed at the beginning of each week for 6 weeks.
  Arms: Exercise and Taping group

SUMMARY:
Neuromuscular exercise and taping are widely used in the rehabilitation of Patellofemoral Pain. The aim of this study was to investigate the effects of corrective kinesio taping applied on patellofemoral joint and foot in addition to a progressive neuromuscular exercise program in women with Patellofemoral Pain on knee pain and muscle strength.

DETAILED DESCRIPTION:
Patellofemoral Pain (PFP) is characterized by pain localized in the peripatellar or retropatellar regions in young and physically active individuals . In patients with PFP, during single-leg squatting, an increase in the valgus of the knee joint due to hip abductor muscle weakness and in the internal rotation of the femur due to weakness of the hip external rotators and abductor muscles are observed. Theoretically it has been shown that faulty hip kinematics can increase lateral loading in the patellofemoral joint. Therefore, conducting exercises to strengthen the extensor, external rotator, and abductor muscles of the hip and lateral flexor muscles of the trunk are an important treatment approaches. Strengthening the quadriceps muscle is a widely used method of treating PFP. Previous studies suggest that hip and trunk exercises prescribed in combination with traditional quadriceps strengthening exercises are effective in reducing pain and improving function in patients with PFP .

In recent years, kinesiotape is one of the widely used methods in the treatment of PFP. The correction of the abnormal patellar displacement, the reduction of the patellofemoral joint reaction forces, and the regulation of the activation of the vastus medialis muscle is provided with patellar taping. Patellar taping is recommended as part of evidence-based combined physiotherapy programs in the treatment of PFP . Increased pronation of the subtalar joint and the decrease / flattening of the medial arch height are associated with PFP. Prolonged pronation time is observed in subtalar and midtarsal joints during gait. To correct increased pronation, foot orthoses, low-dye taping and kinesio taping are applied . The effect of kinesiotaping on foot pronation, however, is unclear due to the lack of published studies.

To our knowledge, although patellar taping is applied in patients with PFP no studies have examined the effects of kinesiotaping supporting the medial arch and allowing forefoot and hind foot to move within the normal range. The aim of this study was to investigate the effects of corrective kinesio taping applied on patellofemoral joint and foot in addition to a progressive neuromuscular exercise program in women with Patellofemoral Pain on knee pain and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* In order for them to be included in the study, it was necessary to have patellofemoral pain in at least two of the long-term sitting, climbing and descending stairs / climbing activities, squatting, running and jumping, and these pains had to continue for at least six months.

Exclusion Criteria:

* Patients with other knee pathologies and knee joint surgery were excluded in the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2015-12-20 (Actual)

PRIMARY OUTCOMES:
Change from Visual Analogue Pain Scale score at 6th. weeks and 12th. weeks | before and after treatment (12 sessions, 6th. and 12th. weeks)]
  The knee pain of the patients during stair descending and ascending were evaluated with the Visual Analogue Pain Scale (VAS). The scale is horizontal in the form of a line 10 cm long, starting with "no pain" and ending with "excruciating pain". The pain was measured and recorded as "cm" between the point marked with no onset .
Change from isokinetic muscle strength of the hamstring and quadriceps femoris muscles at 6th. weeks and 12th. weeks | before and after treatment (12 sessions, 6th. and 12th. weeks)]
  Isokinetic dynamometer (Isomed 2000. D&R. Ferstl GmbH, Germany) was used to evaluate the isokinetic muscle strength of the hamstring and quadriceps femoris muscles. Patients were fixed to the chair with trunk, pelvis, and thigh straps with the back of the seat 70° upright. Concentric peak torque / weight (Nm / kg) at 180° / sec (10 repetitions) after 4 repetitive warm-ups at 180° / sec, in the range of 45 °-90° flexion values were measured, respectively .

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Balcı, Principal Investigator — Muğla Sıtkı Koçman University; Rabia Tugba Kilic, Study Director — Ankara Yildirim Beyazıt University; Volga Bayrakci Tunay, Study Chair — Hacettepe University
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Loudon JK, Wiesner D, Goist-Foley HL, Asjes C, Loudon KL. Intrarater Reliability of Functional Performance Tests for Subjects With Patellofemoral Pain Syndrome. J Athl Train. 2002 Sep;37(3):256-261. PMID 12937582
- [Background] Colado JC, Garcia-Masso X, Triplett NT, Calatayud J, Flandez J, Behm D, Rogers ME. Construct and concurrent validation of a new resistance intensity scale for exercise with thera-band(R) elastic bands. J Sports Sci Med. 2014 Dec 1;13(4):758-66. eCollection 2014 Dec. PMID 25435767
- [Background] Aguilar MB, Abian-Vicen J, Halstead J, Gijon-Nogueron G. Effectiveness of neuromuscular taping on pronated foot posture and walking plantar pressures in amateur runners. J Sci Med Sport. 2016 Apr;19(4):348-53. doi: 10.1016/j.jsams.2015.04.004. Epub 2015 Apr 24. PMID 25956688
- [Background] Baldon Rde M, Serrao FV, Scattone Silva R, Piva SR. Effects of functional stabilization training on pain, function, and lower extremity biomechanics in women with patellofemoral pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):240-251, A1-A8. doi: 10.2519/jospt.2014.4940. Epub 2014 Feb 25. PMID 24568258